CLINICAL TRIAL: NCT00957827
Title: Prophylactic Use of Antibiotics for Through and Through Lacerations of the Lip
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough subject enrolled
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 809859
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Through-and-through Lip Lacerations
MeSH Terms: interventions — Cephalexin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- keflex (Experimental): keflex 500mg twice a day for five days
  Interventions: Drug: keflex
- placebo (Placebo Comparator): placebo 500mg twice a day for five days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: keflex — keflex 500 mg BID 5 days
  Other Names: cephalexin
  Arms: keflex
Drug: placebo — placebo BID for five days
  Arms: placebo

SUMMARY:
Facial lacerations are a commonly encountered problem in the emergency department. Despite this, few original articles have been written concerning the management of lacerations of the lip which communicate with the oral cavity. Specifically, no study has been able to definitively show whether the use of antibiotics for these wounds decreases the infection rate. These cutaneous wounds are a unique type of laceration because they are continuously contaminated with oropharyngeal flora. Contaminated wounds result in larger, less cosmetic scars. Scars which involve the face have been shown to have a negative psychological impact. In this study, the investigators aim to determine whether the use of antibiotics decrease the rate of infection in lacerations of the lip which communicate with the oral cavity. Patients will be randomized to one of two currently practiced therapies. Patients will receive either cephalexin or no treatment following the repair of their through-and-through lip lacerations to determine whether antibiotics decrease the infection rate in these wounds.

DETAILED DESCRIPTION:
Facial lacerations are commonly encountered problem in trauma and emergency room patients. Soft tissue trauma of the face can cause significant psychological impact. Wound care and the need to minimize scarring is particularly important in this region. There have been many studies evaluating the management of soft tissue injuries in general. For example, simple lacerations of the hand do not benefit from antibiotic therapy. The need for antibiotics for full thickness lacerations of the lip, however, has received little attention. Full thickness lacerations of the lip are defined as wounds that violate the mucosa, underlying muscle and skin (i.e through-and through lacerations). These oral-cutaneous injuries constitute a unique type of injury in that the laceration exposes the skin and underlying soft tissue to microbes of the oral pharynx that are normally encountered only by intact oral mucosa. This represents a uniquely different flora from that typically seen in simple skin lacerations. Because these are contaminated wound, there may be an increased risk for infection and an increased need for prophylactic antibiotics. Currently, there is no consensus on the prophylactic treatment of oral-cutaneous wounds with many physicians prescribing oral antibiotics, others utilizing topical antibacterials, and still others treating with local wound care.

A review of the literature found only four original articles addressing the topic of oral antibiotic prophylaxis. Two of these four original articles suffer serious methodological flaws. The first, published in 1965, was a prospective observational study which was neither blinded, nor specified the type or duration of antibiotic therapy. Despite these flaws, the study demonstrated a non-significant trend toward benefit with antibiotics. Of interest, the author noted all wounds older than 24 hours not treated with antibiotics became infected.

The second article, published in 1970 by Paterson et. was a prospective randomized trial, though the type and duration of antibiotic treatment in the intervention arm was left to the discretion of the treating clinician. The author combined both mucosal only oral lacerations and oral-cutaneous wounds. Wound infection was deemed to be present in 18.5% of patients treated with antibiotics versus 4.3% of those receiving no treatment (RR = 4.32, 95% CI = 1.30 to 14.31). None of the patients with mucosa-only wounds developed wound infections; all infections were seen in patients with "through-and-through" lacerations. Despite this, the authors concluded that the role of prophylactic antibiotics is questionable in preventing local infection.

The third article was a prospective, randomized study in the pediatric population evaluating all intra-oral lacerations. In this study 4.3% of patients treated with prophylactic penicillin had evidence of wound infection at follow-up, versus 8.5% of patients in the control arm (RR = 0.51, 95% CI = 0.10 to 2.65). The authors conclude that given the low background rate of infection in this study (8.5%), their study was markedly underpowered, and severely limited their ability to make any conclusions regarding the efficacy of prophylactic antibiotics.

Finally, in 1989, Steele et al. randomized 62 adult patients presenting within 24 hours of injury to a single emergency department with full-thickness intraoral or "through-and-through" lacerations to either treatment with oral antibiotics (penicillin VK for 5 days) or placebo therapy. Among patients treated with penicillin prophylaxis, 6.7% developed wound infection versus 18.8% in the placebo group (RR = 0.36, 95% CI = 0.08 to 1.63). In a subgroup analysis of patients who were perfectly compliant with therapy by pill counts, there were no infections in the penicillin arm versus 17.9% in the placebo arm (p = 0.054 using two-tailed Fisher exact test). The authors alternatively reported this as a statistically significant finding, using a one-tailed Fisher exact test, which yields a p value of 0.027. Furthermore, in subgroup analysis of "through-and-though" lacerations, 7% (1 out of 14) versus 27% (4 out of 15) of patients developed wound infection in the treatment and placebo groups, respectively (RR = 0.27, 95% CI = 0.03 to 2.12). Overall the authors conclude that while they cannot conclusively recommend prophylactic penicillin for adults with intraoral lacerations treated within 24 hours of injury, though there may be a trend towards benefit 9. They also suggest that patients with "through-and-through" wounds may benefit proportionally more from prophylaxis.

Despite the authors' inability to make conclusive recommendations from the available data, many textbooks cite these references and recommend the routine use of antibiotics for oral-cutaneous wounds. Many other text books, on the other hand, do not address this topic at all. Our study aims to answer the question of whether or not antibiotics reduce wound infection rates in through-and-through lacerations of the lip with a dedicated antibiotic regimen evaluated prospectively.

The type of antibiotic used to prophylactically treat oral-cutaneous wounds also remains controversial among clinicians. Previous studies have utilized penicillin V K. Penicillin, however, does not fully cover the flora typically cultured in infected oral-cutaneous wounds. Cephalexin is well described in the literature as an appropriate choice for oropharyngeal infections and has appropriate skin flora coverage, thereby, making it an ideal antibiotic for the prophylaxis of oral-cutaneous wounds.

Current practice concerning the use of antibiotics for oral-cutaneous wounds varies greatly. Many textbooks either do not address the topic or cite inconclusive evidence. A thorough search of the literature revealed only four original articles. No article was able to produce significant results and the trends and recommendations were mixed. Currently, there is no consensus regarding the treatment of oral cutaneous wounds and patients are treated with oral antibiotics, or local wound care depending on the treating physician's preference. It is important to determine the best treatment protocol for these unique wounds.

ELIGIBILITY:
Inclusion Criteria:

* any individual who presents with a through-and-through laceration of the lip within twenty-four hours of injury

Exclusion Criteria:

* patients less than eighteen years of age
* pregnancy
* currently taking antibiotics
* animal or human bites
* wounds greater than 24 hours old
* diabetic patients
* immune compromised patients
* patients who require antibiotics for other sustained injuries
* patients with an allergy to penicillin or cephalosporin will be excluded if randomized to the cephalexin treatment group

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Sims, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hopital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: low enrollment and data not analyzed, patient lost to follow-up.
Period: Overall Study
Arm/Group | Keflex | Placebo
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Keflex | Placebo | Total
Number analyzed (Participants) | 02 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Infection
Description: Presence or absence of infection
Time Frame: one week
Population: Not evaluated due to low enrollment/This should be reflected in all data fields
Arm/Group | Keflex | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: one year
Description: No adverse events
Arm/Group | Keflex | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Study terminated secondary to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No